CLINICAL TRIAL: NCT03893851
Title: Reducing Violent Discipline in School Settings Using Interaction Competencies With Children for Teachers (ICC-T): A Cluster Randomized Controlled Trial in Tanzanian Public Primary Schools
Brief Title: Preventing Violence by Teachers
Acronym: ICC-T_Tz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bielefeld University (Other)
Responsible Party: Principal Investigator, Tobias Hecker, PhD, Resarch Group Leader, Bielefeld University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: ICC-T-Primary-Tz-2019
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Violence by Teachers
Keywords: violence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICC-T (Experimental): Interactions Competencies with Children - for Teachers (ICC-T) 5.5 days with 8 hours of training for teachers. Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting
  Interventions: Behavioral: Interactions Competencies with Children - for Teachers (ICC-T)
- Control (No Intervention): The control schools do not receive any intervention

INTERVENTIONS:
Behavioral: Interactions Competencies with Children - for Teachers (ICC-T) — Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting.
  Arms: ICC-T

SUMMARY:
Brief Summary:

Violence against children is regarded as a key contributor to poverty and damages lifetime prospects for children in disadvantaged communities. However, physical violence is legally accepted as a disciplinary measure in schools in 68 states worldwide. For example, in Tanzania, corporal punishment is still lawful at school. It is thus not surprising that recently very high rates of violence (~90%) were found at secondary schools. For children of primary school age, no such information is available from representative samples to date.

Moreover, in recent studies teachers often report having to resort to violent disciplinary methods referring to a lack of nonviolent disciplinary alternatives . However, only few interventions that aim at equipping teachers with non-violent action alternatives in Sub-Saharan Africa have been implemented, and even fewer have been scientifically evaluated.

Thus, in this study the investigators will implement and assess the efficacy of an intervention aimed at reducing the use of harsh and violent disciplinary measures in schools. Interaction Competencies with Children - for Teacher (ICC-T) aims to enable teachers to use non-violent disciplinary measures and to strengthen their competencies in non-violent interactions. Previously its feasibility and efficacy were proven in secondary schools in Tanzania. The present study aims to adapt ICC-T to, and evaluate its efficacy on, primary school level. The training is expected to improve the teacher-student relationships, change teacher's attitudes towards corporal punishment and their use of violent disciplinary measures.

DETAILED DESCRIPTION:
Sampling will be based on a matched cluster randomized controlled trial design. Study participants (i.e. students, teachers) will be recruited from 6 regions in Tanzania. In each region two primary schools from different districts will be included. From each school 80 pupils and minimum 20 teachers will be recruited. The final sample will comprise 960 pupils in the age-range between 9 and 12 years and at least 240 teachers from 12 different primary schools.

From each region one primary schools will be randomly allocated to the intervention group (that will receive the ICC-T intervention training) and the control group (that will receive no training). The study will have two data assessment points: baseline assessment prior to the intervention and follow-up assessment three months after the intervention. In addition, feasibility data will be assessed in the intervention group at the beginning and the end of the intervention.

Study measures will cover the following topics: socio-demographic data, common disciplinary measure used at school, attitudes towards violent discipline measures, students' mental health problems.

ELIGIBILITY:
Inclusion Criteria:

* • Written informed consent (if underaged by parents & minors)

Exclusion Criteria:

* • Acute drug or alcohol intoxication

  * Acute psychotic disorder

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change of teachers' use of emotional and physical violence | - The CTS will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention).
  - The Conflict Tactics Scale (CTS) will be used to assess teachers' use of emotional and physical violent discipline measures against students. Higher scores indicate higher levels of violence that is used by teachers. We hypothesize a stronger change of the use of violence in the intervention group compared to the control group.
Change of student's exposure to emotional and physical violence by teachers | - The CTS will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention
  - The Conflict Tactics Scale (CTS) will assess the students' self-reported experiences of emotional and physical violence by teachers at school. Higher scores indicate higher levels of violence that is used by teachers. We hypothesize a stronger change of exposure to violence in the intervention group compared to the control group.

SECONDARY OUTCOMES:
Change of student's mental health | - The SDQ will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  - The Strength and Difficulties Questionnaire (SDQ) will assess students' internalizing and externalizing problems. Higher scores indicate higher levels of students' mental health problems. We hypothesize a stronger change of mental health problems in the intervention group compared to the control group.
Change of teachers' attitudes towards emotional and physical violence | - The adapted version of CTS will be used at T 1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  - Teacher's attitudes towards emotional and physical violence will be assessed with an adapted version of the Conflict Tactic Scale (CTS). Higher scores indicate higher levels of positive attitudes towards violence. We hypothesize a stronger change of positive attitudes towards violence in the intervention group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hecker, PhD, Study Chair — Bielefeld University
Locations (1):
- Dar es Salaam University College of Education, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masath FB, Mattonet K, Hermenau K, Nkuba M, Hecker T. Reducing Violent Discipline by Teachers: a Matched Cluster-Randomized Controlled Trial in Tanzanian Public Primary Schools. Prev Sci. 2023 Jul;24(5):999-1010. doi: 10.1007/s11121-023-01550-0. Epub 2023 May 26. PMID 37233888
- [Derived] Masath FB, Hermenau K, Nkuba M, Hecker T. Reducing violent discipline by teachers using Interaction Competencies with Children for Teachers (ICC-T): study protocol for a matched cluster randomized controlled trial in Tanzanian public primary schools. Trials. 2020 Jan 2;21(1):4. doi: 10.1186/s13063-019-3828-z. PMID 31898516